CLINICAL TRIAL: NCT01445080
Title: A Phase I/II Study of the Raf Kinase and Receptor Tyrosine Kinase Inhibitor Sorafenib (BAY 43-9006, NSC# 724772) in Children With Refractory Solid Tumors or Refractory Leukemias
Brief Title: Sorafenib in Treating Young Patients With Relapsed or Refractory Solid Tumors or Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00358; NCI-2009-00358 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 06-C-0233; CDR0000483040; COG-ADVL0413; NCI-06-C-0233; 060233; ADVL0413; ADVL0413 (Other: COG Phase I Consortium); ADVL0413 (Other: CTEP); U01CA097452 (NIH); NCT00343694 (obsolete NCT alias); NCT01648413 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Blastic Phase; Childhood Acute Promyelocytic Leukemia With PML-RARA; Childhood Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Childhood Solid Neoplasm; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Juvenile Myelomonocytic Leukemia; Philadelphia Chromosome Negative, BCR-ABL1 Positive Chronic Myelogenous Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Disease
MeSH Terms: conditions — Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Juvenile; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sorafenib Tosylate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sorafenib Tosylate — Given orally
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This phase I/II trial is studying the side effects and best dose of sorafenib in treating young patients with relapsed or refractory solid tumors or leukemia. Sorafenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum-tolerated dose (MTD) and recommended phase II dose of sorafenib in pediatric patients with relapsed or refractory solid tumors.

II. Determine whether pediatric patients with relapsed or refractory leukemia can tolerate the MTD of sorafenib for solid tumors.

III. Determine the tolerability, active N-oxide metabolite, pharmacodynamics, and activity of sorafenib a the MTD in a subset of patients with acute myeloid leukemia (AML) and FLT3-ITD mutation.

IV. Determine the toxicities of this drug in these patients. V. Determine the pharmacokinetics of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine, preliminarily, the antitumor activity of this drug within the confines of a phase I trial.

II. Assess the biologic effect of sorafenib on circulating endothelial cells (CEC), circulating CEC precursors (CECP), VEGF, and VEGF-2 in peripheral blood.

III. Assess the gene expression, proteomic profile, and ERK phosphorylation in blasts of patients with refractory leukemia treated with this regimen.

IV. Assess the effect of sorafenib on solid tumor vascularity and tumor blood flow using dynamic contrast-enhanced MRI (DEMRI) in patients with measurable soft tissue tumors.

V. Analyze tumor samples and leukemic blasts for the presence of ras, raf, or FLT3 (leukemias) mutations.

VI. Analyze the plasma inhibitory activity for FLT3 phosphorylation in peripheral blood of patients with AML and FLT3-ITD mutation.

VII. Determine the tolerability, pharmacokinetics of sorafenib and sorafenib?s active N-oxide metabolite, pharmacodynamics, and activity of sorafenib administered at the MTD for refractory leukemias in a subset of patients with AML and FLT3-ITD mutation.

VIII. Analyze the plasma inhibitory activity for FLT3 phosphorylation in peripheral blood samples obtained at the time of PK studies in patients with FLT3-ITD mutation AML.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to diagnosis (malignant solid tumor vs leukemia).

STRATUM I(REFRACTORY SOLID TUMOR PATIENTS): Patients receive oral sorafenib twice daily on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of sorafenib until the maximum-tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT). Once the MTD is determined, up to 6 additional patients under 12 years of age may be treated at the MTD. The MTD dose level is also expanded to enroll up to 6 patients with refractory leukemia.

STRATUM II (REFRACTORY LEUKEMIA PATIENTS): A cohort of 3-6 patients with leukemia receives treatment as in stratum 1 at the MTD determined in stratum 1. If 2 of 3 or 2 of 6 patients experience a DLT at the solid tumor MTD, sorafenib is reduced by one dose level. The leukemia MTD is defined as the dose at which < 1/3 of patients experience DLT during course 1 of treatment.

STRATUM III (ACUTE MYELOID LEUKEMIA AND FLT3-ITD MUTATION PATIENTS): Patients receive sorafenib as in stratum 1 at the MTD determined in stratum 2. Patients undergo blood sample collection for pharmacokinetics, pharmacodynamics (in leukemia blasts only), circulating endothelial cells (CEC), circulating CEC precursors (CECP), VEGF and VEGF-2 , gene expression, proteomic profile, ERK phosphorylation, and FLT3 phosphorylation activity. Tumor tissue samples may also be analyzed for the presence of ras, raf, or FLT3.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Histologically confirmed malignant solid tumor at original diagnosis or relapse

    * Measurable or evaluable disease by CT scan or MRI
  * Histologically confirmed leukemia, including 1 of the following:

    * Acute lymphoblastic leukemia (ALL)

      * Greater than 25% blasts in the bone marrow (M3 bone marrow)
    * Acute myeloid leukemia (AML)

      * Greater than 25% blasts in the bone marrow (M3 bone marrow)
    * AML and FLT3-ITD mutation

      * Patients must have ? 5% blasts in the bone marrow
      * Active extramedullary disease (except leptomeningeal disease) allowed
    * Juvenile myelomonocytic leukemia (JMML) meeting the following criteria:

      * Peripheral blood monocytosis > 1,000/mm^3
      * Blasts (including promonocytes) are < 20% of the WBCs in the blood and of the nucleated bone marrow cells
      * No Philadelphia chromosome (Ph) or BCR/ABL fusion gene
      * Has ? 2 of the following additional diagnostic criteria:

        * Hemoglobin F increased for age
        * Immature granulocytes in the peripheral blood
        * WBC > 10,000/mm^3
        * Clonal chromosomal abnormality (e.g., may be monosomy 7)
        * Sargramostim (GM-CSF) hypersensitivity of myeloid progenitors in vitro
    * Chronic myelogenous leukemia (CML) in blast crisis

      * Greater than 25% blasts in the bone marrow (M3 bone marrow)
      * Patients with Ph-positive CML must be refractory to imatinib mesylate
* Relapsed or refractory disease

  * Patients with acute promyelocytic leukemia (APL) must be refractory to treatment with tretinoin and arsenic trioxide
* Standard curative therapies or therapies proven to prolong survival with an acceptable quality of life do not exist
* Active extramedullary disease, except active leptomeningeal leukemia, allowed
* No brain tumors or known brain metastases
* Karnofsky performance status (PS) 50-100% (for patients > 10 years of age)
* Lansky PS 50-100% (for patients ? 10 years of age)
* Patients with solid tumors must have adequate bone marrow function, as defined by the following:

  * Absolute neutrophil count ? 1,000/mm^3
  * Platelet count ? 75,000/mm^3 (transfusion independent)
  * Hemoglobin ? 8.0 g/dL (red blood cell [RBC] transfusions allowed)
* Patients with leukemia may have abnormal blood counts but must meet the following criteria:

  * Platelet count ? 20,000/mm^3 (platelet transfusions allowed)
  * Hemoglobin ? 8.0 g/L (RBC transfusions allowed)
* Patients with acute myeloid leukemia and FLT3-ITD mutation

  * Platelet count ? 20,000/mm^3
* Lipase and amylase normal
* Creatinine clearance or radioisotope glomerular filtration rate ? 70 mL/min OR creatinine normal based on age as follows:

  * No greater than 0.8 mg/dL (for patients 5 years of age and under)
  * No greater than 1.0 mg/dL (for patients 6-10 years of age)
  * No greater than 1.2 mg/dL (for patients 11-15 years of age)
  * No greater than 1.5 mg/dL (for patients over 15 years of age)
* Patients with solid tumors must meet the following criteria:

  * Bilirubin normal for age
  * ALT normal for age (for the purpose of this study, the upper limit of normal [ULN] for ALT is 45 ?/L)
  * Serum albumin ? 2 g/dL
* Patients with leukemia must meet the following criteria:

  * Bilirubin (sum of conjugated + unconjugated) ? 1.5 times ULN for age
  * ALT ? 5.0 times ULN for age (? 225 ?/L) (for the purpose of this study, the ULN for ALT is 45 ?/L)
  * Serum albumin ? 2 g/dL
* Albumin ? 2 g/dL
* PT, PTT, and INR normal (for patients on prophylactic anticoagulation)
* No evidence of dyspnea at rest
* No exercise intolerance
* Pulse oximetry >94% on room air, if there is clinical indication for determination
* Diastolic blood pressure ? the 95th percentile for age and gender (height included for AML and FLT3-ITD mutation patients)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* Able to swallow tablets
* No evidence of bleeding diathesis
* No other medical condition or situation that would preclude study compliance
* No known Gilbert syndrome
* Fully recovered from prior chemotherapy, immunotherapy, or radiotherapy (for patients with solid tumors)
* Recovered from the non-hematologic toxic effects of all prior therapy (for patients with leukemia)
* Recovered from acute non-hematologic toxic effects of all prior anti-cancer chemotherapy (for patients with AML and FLT3-ITD mutation)
* At least 7 days since prior hematopoietic growth factors
* At least 7 days since prior biologic agents
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 3 months since prior total-body irradiation, craniospinal radiotherapy, or radiation to ? 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiation (e.g., skull, spine, pelvis, ribs)
* At least 3 months since prior stem cell transplantation or rescue (for patients with solid tumors)

  * No evidence of active graft-vs-host disease
* At least 3 months since prior myeloablative therapy followed by bone marrow or stem cell transplantation (for patients with leukemia)
* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) (for patients with solid tumors)

  * At least 24 hours since prior nitrosoureas (for patients with AML and FLT3-ITD mutation)
* At least 2 weeks since prior chemotherapy (for patients with leukemia)
* At least 3 weeks since prior monoclonal antibody therapy
* No prior sorafenib
* No other concurrent investigational drugs
* No other concurrent anticancer agents or therapies, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy

  * Concurrent maintenance-like chemotherapy for patients with AML and FLT3-ITD mutation allowed
* No concurrent administration of any of the following:

  * Cytochrome P450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital)
  * Rifampin
  * Grapefruit juice
  * Hypericum perforatum (St. John wort)
* No concurrent therapeutic anticoagulation

  * Concurrent prophylactic anticoagulation (e.g., low-dose warfarin) of venous or arterial access devices allowed provided the requirements for PT, INR, or PTT are met

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2006-05-30 (Actual); Primary Completion 2012-03-16 (Actual); Study Completion 2012-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, Principal Investigator — COG Phase I Consortium
Locations (25):
- United States (23):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2: Patients receive oral sorafenib 105 mg/m^2 every 12 hours.
- Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2: Patients receive oral sorafenib 130 mg/m^2 every 12 hours.
- Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2; Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2; Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2: Patients receive oral sorafenib 150 mg/m^2 every 12 hours.
- Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2; Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2; PK Cohort Expanded: BAY 43-9006 200 mg/m^2: Patients receive oral sorafenib 200 mg/m^2 every 12 hours.
- Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2: Patients receive oral sorafenib 250 mg/m^2 every 12 hours.
Period: Overall Study
Arm/Group | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2 | PK Cohort Expanded: BAY 43-9006 200 mg/m^2
Started | 7 | 5 | 12 | 8 | 4 | 9 | 2 | 5 | 18
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 5 | 12 | 8 | 4 | 9 | 2 | 5 | 18
Not completed — Adverse Event | 5 | 3 | 11 | 6 | 2 | 3 | 0 | 3 | 10
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Ineligible/Inevaluable | 1 | 2 | 0 | 1 | 2 | 3 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2 | PK Cohort Expanded: BAY 43-9006 200 mg/m^2 | Total
Number analyzed (Participants) | 7 | 5 | 12 | 8 | 4 | 9 | 2 | 5 | 18 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 11 | 6 | 4 | 8 | 2 | 5 | 15 | 60
  Between 18 and 65 years | 3 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 3 | 10
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 17 [9 to 21] | 16 [14 to 18] | 13.5 [5 to 21] | 13.5 [6 to 21] | 11.5 [6 to 14] | 13 [6 to 19] | 10.5 [6 to 15] | 12 [4 to 18] | 14.5 [5 to 21] | 14 [4 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 9 | 3 | 1 | 1 | 0 | 0 | 4 | 23
  Male | 3 | 4 | 3 | 5 | 3 | 8 | 2 | 5 | 14 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 3 | 0 | 2 | 1 | 0 | 1 | 2 | 11
  Not Hispanic or Latino | 5 | 4 | 8 | 8 | 1 | 8 | 2 | 4 | 16 | 56
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 3 | 7
  White | 6 | 2 | 10 | 5 | 2 | 8 | 1 | 3 | 15 | 52
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-related Dose Limiting Toxicity in Cycle 1 by Dose Level
Description: Number of patients with treatment-related dose limiting toxicities in cycle 1, as defined by study protocol, stratified by dose level.
Time Frame: Up to 28 days
Population: There were 55 evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2 | PK Cohort Expanded: BAY 43-9006 200 mg/m^2
Number analyzed (Participants) | 6 | 3 | 12 | 7 | 2 | 6 | 2 | 5 | 12
Participants | 0 | 0 | 5 | 1 | 2 | 0 | 2 | 0 | 3

2. Primary Outcome: Number of Patients With Treatment-related Adverse Events
Description: Number of patients with treatment-related adverse events stratified by dose level through study completion.
Time Frame: Up to 2 years
Population: There were 55 evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2 | PK Cohort Expanded: BAY 43-9006 200 mg/m^2
Number analyzed (Participants) | 7 | 5 | 12 | 8 | 4 | 9 | 2 | 5 | 18
Participants | 6 | 3 | 12 | 7 | 2 | 6 | 2 | 5 | 12

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Sorafenib
Description: Area under the plasma concentration versus time curve (AUC) of sorefenib administered orally as tablets, BID approximately every 12 hours for cycles of 28 days with no rest period between cycles to children with refractory solid tumors or leukemias.
Time Frame: During cycle 1 or cycle 2 after at least 14 consecutive days of sorafenib administration Pre-dose, 0.5, 1, 2, 3, 5, 8 hours post dose
Population: Pharmacokinetic (PK) studies were completed for stratums I and II. Summary statistics for PK analysis was performed regardless of dose level as pre-specified in the protocol. PK was not performed in stratum III
Measure: Mean (Full Range); unit: µg•h/ml
Groups:
- STRATUM I (REFRACTORY SOLID TUMOR): Patients receive oral sorafenib twice daily on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of sorafenib until the maximum-tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT). Once the MTD is determined, up to 6 additional patients under 12 years of age may be treated at the MTD. The MTD dose level is also expanded to enroll up to 6 patients with refractory leukemia.
- STRATUM II (REFRACTORY LEUKEMIA): A cohort of 3-6 patients with leukemia receives treatment as in stratum 1 at the MTD determined in stratum 1. If 2 of 3 or 2 of 6 patients experience a DLT at the solid tumor MTD, sorafenib is reduced by one dose level. The leukemia MTD is defined as the dose at which < 1/3 of patients experience DLT during course 1 of treatment
Arm/Group | STRATUM I (REFRACTORY SOLID TUMOR) | STRATUM II (REFRACTORY LEUKEMIA)
Number analyzed (Participants) | 29 | 5
µg•h/ml | 38.66 [2.54 to 104.61] | 50.03 [20.25 to 97.78]

4. Primary Outcome: Clearance (Cl) of Sorafenib
Description: Clearance of sorefenib administered orally as tablets, BID approximately every 12 hours for cycles of 28 days with no rest period between cycles to children with refractory solid tumors or leukemias.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Full Range); unit: mL/min/m^2
Groups:
- STARTUM I (REFRACTORY SOLID TUMORS): Patients receive oral sorafenib twice daily on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of sorafenib until the maximum-tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT). Once the MTD is determined, up to 6 additional patients under 12 years of age may be treated at the MTD. The MTD dose level is also expanded to enroll up to 6 patients with refractory leukemia.
Arm/Group | STARTUM I (REFRACTORY SOLID TUMORS) | STRATUM II (REFRACTORY LEUKEMIA)
Number analyzed (Participants) | 13 | 4
mL/min/m^2 | 57.2 [19.2 to 130] | 72.6 [24.4 to 121]

5. Primary Outcome: Half-life of Sorafenib
Description: Half-life of sorefenib administered orally as tablets, BID approximately every 12 hours for cycles of 28 days with no rest period between cycles to children with refractory solid tumors or leukemias.
Time Frame: as for outcome 3
Population: Data was and never will be collected
Groups:
- STRATUM I (REFRACTORY SOLID TUMOR: Patients receive oral sorafenib twice daily on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of sorafenib until the maximum-tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT). Once the MTD is determined, up to 6 additional patients under 12 years of age may be treated at the MTD. The MTD dose level is also expanded to enroll up to 6 patients with refractory leukemia.
Arm/Group | STRATUM I (REFRACTORY SOLID TUMOR | STRATUM II (REFRACTORY LEUKEMIA)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Maximum Serum Concentration (Cmax) of Sorafenib
Description: Maximum serum concentration (Cmax) of sorefenib administered orally as tablets, BID approximately every 12 hours for cycles of 28 days with no rest period between cycles to children with refractory solid tumors or leukemias.
Time Frame: as for outcome 3
Population: Data was not collected for patients from Part A:130 mg/m^2
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 | PK Cohort Expanded: BAY 43-9006 200 mg/m^2
Number analyzed (Participants) | 4 | 9 | 4 | 1 | 4 | 1 | 11
µg/ml | 0.71 (0.53) | 1.88 (1.55) | 1.98 (1.25) | 1.80 (0) | 5.97 (4.45) | 5.02 (0) | 7.95 (.43)

7. Primary Outcome: Number of Patients With Treatment-related Dose Limiting Toxicities in Later Cycles by Dose Level
Description: Number of patients with treatment-related dose limiting toxicities in later cycles, as defined by study protocol, stratified by dose level.
Time Frame: Up to 2 years
Population: There were 55 evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2 | PK Cohort Expanded: BAY 43-9006 200 mg/m^2
Number analyzed (Participants) | 6 | 3 | 12 | 7 | 2 | 6 | 2 | 5 | 12
Participants | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2

8. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Sorafenib
Description: Area under the plasma concentration versus time curve (AUC) of sorefenib administered orally as tablets, BID approximately every 12 hours for cycles of 28 days with no rest period between cycles to children with AML and FLT3-ITD mutation.
Time Frame: 8 hours post dose on day 1 of cycle 1
Population: Data was and never will be collected
Groups:
- STRATUM III (ACUTE MYELOID LEUKEMIA AND FLT3-ITD MUTATION): Patients receive sorafenib as in stratum 1 at the MTD determined in stratum 2. Patients undergo blood sample collection for pharmacokinetics, pharmacodynamics (in leukemia blasts only), circulating endothelial cells (CEC), circulating CEC precursors (CECP), VEGF and VEGF-2 , gene expression, proteomic profile, ERK phosphorylation, and FLT3 phosphorylation activity. Tumor tissue samples may also be analyzed for the presence of ras, raf, or FLT3.
Arm/Group | STRATUM III (ACUTE MYELOID LEUKEMIA AND FLT3-ITD MUTATION)
Number analyzed (Participants) | 0

9. Primary Outcome: Clearance (Cl) of Sorafenib
Description: Clearance of Sorefenib administered orally as tablets, BID approximately every 12 hours for cycles of 28 days with no rest period between cycles to children with AML and FLT3-ITD mutation.
Time Frame: 8 hours post dose on day 1 of cycle 1
Population: Data was and never will be collected
Arm/Group | STRATUM III (ACUTE MYELOID LEUKEMIA AND FLT3-ITD MUTATION)
Number analyzed (Participants) | 0

10. Primary Outcome: Half-life of Sorafenib
Description: Half-life of sorefenib administered orally as tablets, BID approximately every 12 hours for cycles of 28 days with no rest period between cycles to children with AML and FLT3-ITD mutation.
Time Frame: 8 hours post dose on day 1 of cycle 1
Population: Data was and never will be collected
Arm/Group | STRATUM III (ACUTE MYELOID LEUKEMIA AND FLT3-ITD MUTATION)
Number analyzed (Participants) | 0

11. Primary Outcome: Volume of Distribution at Steady State (Vss) of Sorafenib
Description: Volume of distribution at steady state (Vss) of sorefenib administered orally as tablets, BID approximately every 12 hours for cycles of 28 days with no rest period between cycles to children with refractory solid tumors, leukemia, or AML and FLT3-ITD mutation.
Time Frame: 8 hours post dose on day 1 of cycle 1
Population: Data was and never will be collected
Arm/Group | STRATUM I (REFRACTORY SOLID TUMOR | STRATUM II (REFRACTORY LEUKEMIA) | STRATUM III (ACUTE MYELOID LEUKEMIA AND FLT3-ITD MUTATION)
Number analyzed (Participants) | 0 | 0 | 0

12. Primary Outcome: Maximum Serum Concentration (Cmax) of Sorafenib
Description: Maximum serum concentration (Cmax) of Sorefenib administered orally as tablets, BID approximately every 12 hours for cycles of 28 days with no rest period between cycles to children with AML and FLT3-ITD mutation.
Time Frame: 8 hours post dose on day 1 of cycle 1
Population: Data was and never will be collected
Arm/Group | STRATUM III (ACUTE MYELOID LEUKEMIA AND FLT3-ITD MUTATION)
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Patients Who Respond Using RECIST Criteria
Description: Frequency (%) of patients with Partial Response (PR) or Complete Response (CR) using the RECIST criteria by study part and dose level
Time Frame: Up to 2 years
Population: There were 55 evaluable patients
Measure: Number; unit: participants
Arm/Group | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2 | PK Cohort Expanded: BAY 43-9006 200 mg/m^2
Number analyzed (Participants) | 6 | 3 | 12 | 7 | 2 | 6 | 2 | 5 | 12
participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0

14. Secondary Outcome: Mean Concentration of VEGF2
Description: Mean concentration of VEGF2 in peripheral blood sample.
Time Frame: 28 days
Population: Data were not collected for Part A: 250 mg/m^2, Part B:150 mg/m^2, Part B: 200 mg/m^2, and Part C:150 mg/m^2
Measure: Mean (Standard Deviation); unit: cells/ml
Arm/Group | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 | PK Cohort Expanded: BAY 43-9006 200 mg/m^2
Number analyzed (Participants) | 4 | 2 | 5 | 3 | 4
cells/ml | 2650 (2243.49) | 247.5 (258.09) | 3531.5 (4775.11) | 430 (324.50) | 100 (124.90)

15. Secondary Outcome: Pharmacodynamics (PD) Blood Flow Part C
Description: Pharmacodynamics: tumor blood flow in patients with AML and FLT3-ITD mutation using dynamic contrast enhanced MRI (DEMRI) (Part C).
Time Frame: 1 week prior to enrollment, then every 28 days
Population: This data were not and will never be collected
Arm/Group | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Patients With DEMRI
Description: Assess effect on tumor blood flow via DEMRI in patients with measurable soft tissue tumors.
Time Frame: Up to 2 years
Population: There were 55 evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2 | PK Cohort Expanded: BAY 43-9006 200 mg/m^2
Number analyzed (Participants) | 6 | 3 | 12 | 7 | 2 | 6 | 2 | 5 | 12
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Leukemia Mutations
Description: Analyze tumor samples and leukemic blasts from patients entered on this study for the presence of ras, raf, or FLT3 (leukemia) mutations.
Time Frame: 1 week prior to enrollment
Population: This data were not and will never be collected
Arm/Group | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2
Number analyzed (Participants) | 0

18. Secondary Outcome: Plasma Inhibitory Activity (PIA)
Description: Analyze the plasma inhibitory activity (PIA) for FLT3 phosphorylation in peripheral blood samples obtained at the time of PK studies in patients with FLT3-ITD mutation AML (Part C).
Time Frame: 1 week prior to enrollment and then every 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Groups:
- Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2; Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2: Patients receive oral sorafenib 250 mg/m^2 every 12 hours.
Arm/Group | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2 | PK Cohort Expanded: BAY 43-9006 200 mg/m^2
All-Cause Mortality (participants affected / at risk) | 7/7 | 5/5 | 12/12 | 8/8 | 2/4 | 9/9 | 2/2 | 5/5 | 18/18
Serious Adverse Events (participants affected / at risk) | 7/7 | 5/5 | 12/12 | 8/8 | 2/4 | 9/9 | 2/2 | 5/5 | 18/18
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5 | 12/12 | 8/8 | 2/4 | 9/9 | 2/2 | 5/5 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 (N=7) | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 (N=5) | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 (N=12) | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 (N=8) | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 (N=4) | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 (N=9) | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 (N=2) | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2 (N=5) | PK Cohort Expanded: BAY 43-9006 200 mg/m^2 (N=18)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 0 | 1 | 6 | 2 | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Edema face (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 2 | 0
Fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 1 | 2 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 0
INR increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 2 | 2 | 1 | 3 | 2 | 5 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 4 | 5
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 8 | 1 | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden death NOS (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 2 | 0 | 1 | 2 | 0 | 3 | 1 | 5 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Refractory Solid Tumors: BAY 43-9006 105 mg/m^2 (N=7) | Part A: Refractory Solid Tumors: BAY 43-9006 130 mg/m^2 (N=5) | Part A: Refractory Solid Tumors: BAY 43-9006 150 mg/m^2 (N=12) | Part A: Refractory Solid Tumors: BAY 43-9006 200 mg/m^2 (N=8) | Part A: Refractory Solid Tumors: BAY 43-9006 250 mg/m^2 (N=4) | Part B: Refractory Leukemia: BAY 43-9006 150 mg/m^2 (N=9) | Part B: Refractory Leukemia: BAY 43-9006 200 mg/m^2 (N=2) | Part C: Refractory AML With FLT3-ITD Mutation:150 mg/m^2 (N=5) | PK Cohort Expanded: BAY 43-9006 200 mg/m^2 (N=18)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 3 | 1 | 1 | 4 | 1 | 2 | 3
Acidosis (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0 | 1 | 2 | 0 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 1 | 0 | 0 | 5 | 2 | 2 | 2
Agitation (Psychiatric disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 5 | 2 | 2 | 4 | 2 | 4 | 10
Alkaline phosphatase increased (Investigations) | 2 | 0 | 3 | 0 | 1 | 1 | 0 | 1 | 2
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 3
Anal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 5 | 2 | 1 | 5 | 1 | 3 | 7
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 2 | 4 | 1 | 2 | 8
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 8 | 2 | 1 | 6 | 2 | 4 | 10
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2 | 0 | 2 | 0 | 1 | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Blood bilirubin increased (Investigations) | 2 | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 6
Blurred vision (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0 | 3 | 0 | 1 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0
Cholesterol high (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 0 | 2 | 1 | 0 | 6 | 0 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 4 | 4
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 6 | 5 | 2 | 6 | 0 | 0 | 10
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 3 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 0 | 3 | 0 | 3 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Edema face (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 6 | 4 | 2 | 8 | 1 | 5 | 11
Fever (General disorders) | 2 | 0 | 4 | 1 | 0 | 1 | 1 | 2 | 5
Fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flashing lights (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
GGT increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 1 | 3 | 2 | 0 | 4 | 2 | 3 | 2
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3 | 5 | 2 | 1 | 8 | 2 | 3 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 2 | 0 | 2 | 1 | 1 | 2
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 3 | 2 | 5 | 1 | 2 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 6 | 2 | 2 | 6 | 2 | 4 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 6 | 2 | 2 | 5 | 2 | 4 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 3 | 1 | 7 | 1 | 1 | 5 | 2 | 2 | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 2 | 4 | 2 | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 2 | 1 | 5 | 2 | 2 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1 | 5 | 2 | 2 | 5 | 1 | 1 | 10
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 3 | 1 | 2 | 0
INR increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Investigations - Other, specify (Investigations) | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 2
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 3 | 2 | 1 | 5 | 0 | 1 | 9
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 4 | 1 | 3 | 4
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 5 | 4 | 1 | 6 | 1 | 3 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1 | 3 | 3 | 0 | 1 | 0 | 1 | 8
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 2 | 1 | 3 | 0 | 1 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2 | 1 | 1 | 1 | 3 | 2
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 4 | 0 | 3 | 3 | 1 | 0 | 0 | 3 | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0 | 3 | 1 | 0 | 3 | 1 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1 | 5 | 5 | 1 | 5 | 0 | 4 | 8
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Serum amylase increased (Investigations) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 4
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 5 | 0 | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 5 | 3 | 1 | 6 | 1 | 4 | 7
Weight gain (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight loss (Investigations) | 1 | 0 | 1 | 3 | 1 | 4 | 0 | 1 | 3
White blood cell decreased (Investigations) | 4 | 1 | 6 | 3 | 1 | 2 | 1 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less